CLINICAL TRIAL: NCT02734381
Title: Prevalence of Presenting Diseases for Elderly Patients Admitted to Emergency Department
Status: Completed | Type: Observational
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Umut Gulacti, Principal Investigator, Adiyaman University Research Hospital
Other Study IDs: ADYU 5
Record Dates: First submitted 2016-04-07; First posted 2016-04-12 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Geriatric Disorder
Keywords: elderly patients; prevalence; emergency department use; main presenting disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Elderly patients — Elderly patients who visited the Emergency Department

SUMMARY:
The number of elderly patients admitted to the Emergency Department (ED) is dramatically increasing.

DETAILED DESCRIPTION:
The number of elderly patients admitted to the Emergency Department (ED) is dramatically increasing. Most emergency physicians have not been trained in specific geriatric approaches, and many report being less comfortable when dealing with older patients. Aim of this study is the investigation the most common conditions affecting older patients in the ED.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients who visited the Emergency Department

Exclusion Criteria:

* Patients below 65 years of age
* Patients with missing data in medical records

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients who visited the Emergency Department of Adiyaman University of Training and Research Hospital between 1 January 2015 and 1 December 2015.
Sampling Method: Non-Probability Sample
Enrollment: 36369 (Actual)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The use of Emergency department by Syrian refugees | one year
  The emergency department visits of elderly patients by data obtained from medical records

CONTACTS AND LOCATIONS:
Overall Officials: Umut Gulacti, Principal Investigator — Adiyaman University of Medical Faculty
Locations (1):
- Adiyaman University Research Hospital, Adıyaman, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Geurts J, Palatnick W, Strome T, Sutherland KA, Weldon E. Frequent users of an inner-city emergency department. CJEM. 2012 Sep;14(5):306-13. doi: 10.2310/8000.2012.120670. PMID 22967698
- [Background] Samaras N, Chevalley T, Samaras D, Gold G. Older patients in the emergency department: a review. Ann Emerg Med. 2010 Sep;56(3):261-9. doi: 10.1016/j.annemergmed.2010.04.015. PMID 20619500